CLINICAL TRIAL: NCT07195435
Title: The Effect of Peer Education on Genital Hygiene Behaviors and Self-Care Power in Adolescent Girls
Brief Title: Peer Education on Genital Hygiene and Self-Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Fatma Keskin Töre, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/21
Record Dates: First submitted 2025-09-15; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Genital Hygiene Behaviors; Self-Care
Keywords: genital hygiene; Self-Care; Peer Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genital Hygiene Training: (Experimental)
  Interventions: Behavioral: Genital Hygiene Education
- Control Group (No Intervention): The young girls in the control group will complete a pre-test form consisting of a Personal Information Form, a Genital Hygiene Behavior Scale, and a Self-Care Ability Scale. Four weeks later, in a post-test, the aforementioned scale questions will be asked again.

INTERVENTIONS:
Behavioral: Genital Hygiene Education — Genital Hygiene Training: Young girls who agree to participate will receive two sessions of two hours of genital hygiene training on a predetermined date, as appropriate. Genital hygiene training will be delivered via PowerPoint presentation, and at the end of the training, a training booklet and brochure, developed in accordance with the relevant literature, will be distributed to the participating girls to ensure retention. The training booklet and brochure will be prepared by the researcher based on current literature sources. Expert opinions will be sought from obstetrics and gynecology nursing experts regarding the training content and will be revised as necessary. The content of the training booklet will cover the female internal and external genital organs, the importance of genital infections for women's health, factors affecting genital hygiene, characteristics of normal and abnormal genital discharge, common genital infections, signs and symptoms of genital infection, and pro
  Arms: Genital Hygiene Training:

SUMMARY:
This study was conducted to determine the effects of peer education provided to teenage girls on genital hygiene behaviors and self-care agency. The study was conducted with a randomized controlled design with a pretest-posttest control group. The study was conducted with female students studying at Kahramanmaraş Sütçü İmam University Technical Sciences Vocational School between October and November 2025. The research population consisted of all female students at the school, and the sample consisted of students who agreed to participate in the study, signed the consent form, and met the inclusion criteria. Data were collected using a "Personal Information Form," a "Genital Hygiene Behaviors Scale," and a "Self-Care Agency Scale." Peer education was administered to the intervention group, while the control group received no training.

DETAILED DESCRIPTION:
Genital infections are the most common cause of hospital admissions for reproductive health. While these infections are treatable and preventable, they can negatively impact women's health due to their complications. Genital infections are among the most preventable diseases, but due to their prevalence and complications, they pose a significant problem for women's health. Genital infections are both preventable and treatable, but they are a major problem frequently encountered among women aged 15-49. Women most frequently present to gynecology clinics with complaints of itching and vaginal discharge. Genital infections cause various complications related to reproductive health. Genital infections can negatively impact a woman's fertility, sexual life, family life, and mental health, impairing her quality of life, and can also lead to social isolation. Literature reports that approximately one million women worldwide experience genital infections annually, and 75% of them have a history of vaginal infections. Studies conducted in Turkey indicate that women have inadequate/incorrect genital hygiene practices and a low level of awareness.

Factors such as the anatomical structure of the female genital system, inadequate knowledge about preventing genital infections, low socioeconomic status, inadequate/incorrect perineal and menstrual hygiene, not washing hands before and after using the toilet, and not using appropriate underwear contribute to genital infections. The main factor that can be changed in preventing genital infections is deficiencies in genital and menstrual hygiene. Genital hygiene encompasses many different hygiene behaviors necessary to protect the organs in the genital area from infectious agents, maintain body health, and improve functional health conditions. Ensuring genital hygiene is of great importance in protecting and improving women's health. When genital hygiene is not given the necessary attention, the tendency to genital infection increases, and if genital infection is left untreated, a woman's fertility is affected. Therefore, correctly implemented genital hygiene behaviors are the most critical step in preventing genital infections and their consequences. When studies conducted in our country are examined; As a result of lack of knowledge and incorrect practices about genital hygiene behaviors, women are seen to present to outpatient clinics with complaints of genital discharge, and their risk of vaginal infection increases. Therefore, it is emphasized that education focusing on correct genital hygiene habits has the potential to reduce this risk. Nurses, as part of the healthcare system, play a critical role in improving the health behaviors of both individuals and society through the educational seminars they conduct. This type of health education provided to women positively affects not only their personal health but also public health. Studies have shown that education covering correct genital hygiene practices can contribute to women's health, strengthening their self-care ability, physical health, mental health, and social relationships. There are many "self-care" practices that people perform to maintain their health. Genital hygiene care has an important place among these. Good self-care practices positively impact quality of life through factors such as preventing illness, providing a sense of independence and control, and contributing to personal development. However, this relationship can vary from person to person depending on individual experiences. Genital infections reduce individuals' standards of living and negatively affect their self-care ability. Increasing self-care ability, one of the factors that plays a role in preventing genital infections, is crucial. Therefore, this study aimed to examine the effects of peer education provided to young girls on genital hygiene behavior and self-care ability.

Research Type: This is a pretest-posttest randomized controlled trial. The study was conducted with female students studying at Kahramanmaraş Sütçü İmam University Technical Vocational School between the dates of the study.

Research Universe and Sample: The study population consists of female students studying at Kahramanmaraş Sütçü İmam University (KSU) Technical Sciences Vocational School. The study sample will consist of students who were continuing their education between October and November 2025, agreed to participate in the study, signed the consent form, and met the inclusion criteria.

The sample size of the study was calculated based on the findings of the randomized controlled trial by Sabancı Baransel et al. (2024). In this study, a significant increase in the total score of the Genital Hygiene Behaviors Inventory was found in the intervention group, and the difference between the groups at the posttest was found to be large effect size (Cohen's d ≈ 1.0-1.2). In light of these data, a power analysis was conducted for our study using ANCOVA analysis in a pretest-posttest design between two groups (experimental and control) using G*Power 3.1. Based on the criteria of a medium-to-large effect size (Cohen's d = 0.80), 95% confidence level (α = 0.05), and 80% power (1-β = 0.80), a minimum of 30 participants per group was calculated. Considering a possible 20% sample loss, a total of 72 students were targeted, with 36 participants per group.

After receiving ethics committee approval for the study, young girls living at the Kahramanmaraş Onikişubat Girls' Dormitory who meet the inclusion criteria will be informed about the purpose and content of the study upon their first meeting. Participants who meet the inclusion criteria and agree to participate will provide verbal and written consent. Pre-test data will be collected using a 16-question Personal Information Form, a 23-item Genital Hygiene Behaviors Scale, and a 35-item Self-Care Abilities Scale. Administration of these tests takes approximately 15 minutes. Post-test data will be collected four weeks after the pre-test data using the Genital Hygiene Behaviors Scale and the Self-Care Abilities Scale via face-to-face interviews by the researcher.

Randomization KSU-Technical Sciences Vocational School has seven departments. An independent person, not involved in the study, placed cards bearing the names of these seven sections in opaque, sealed envelopes. The researchers randomly selected the envelopes without knowing their contents; the first selected envelope was assigned to the intervention group (genital hygiene education), and the second envelope was assigned to the control group. Thus, randomization was performed at the department level (cluster randomization) in a 1:1 ratio. Students from both departments were listed, and female students who met the inclusion criteria and provided written informed consent were included in the study. Participant recruitment continued until the predetermined sample size was reached. To reduce potential contamination, intervention and control sessions were conducted at different times and/or locations, and the sharing of educational materials between groups was limited.

Data Collection Tools Data will be collected using a Personal Information Form, the Genital Hygiene Behaviors Scale, and the Self-Care Ability Scale.

Personal Information Form Developed by researchers based on literature, the Personal Information Form consists of a total of 16 questions: four questions regarding female students' socio-demographic characteristics (age, grade, income), three questions regarding their dormitory environment (such as number of people in a room, shared toilets and bathrooms), three questions regarding gynecological characteristics (such as history of genital infections, use of sanitary pads), and six questions regarding hygiene habits.

Genital Hygiene Behaviors Scale The scale was developed by Karahan in 2017. The five-point Likert-type scale consists of 23 items. The scale consists of three subscales: "General Hygiene Behaviors," "Menstrual Hygiene," and "Awareness of Abnormal Findings." The scale, which measures women's genital hygiene behaviors, can be scored with a minimum score of 23 and a maximum score of 115. As the score on the scale increases, the rate of women exhibiting correct genital hygiene behavior also increases.

Self-Care Ability Scale Developed by Kearney and Fleischer in 1979 to determine individuals' self-care abilities, the scale's validity and reliability in Turkish were conducted by Nahcivan in 1993. Each statement on the thirty-five-item scale is a 5-point Likert-type scale ranging from 0 to 4. "Doesn't describe me at all" receives 0 points, "Doesn't describe me very much" receives 1 point, "I have no idea" receives 2 points, "Describes me a little" receives 3 points, and "Describes me a lot" receives 4 points. Eight statements on the scale (3, 6, 9, 13, 19, 22, 26, and 31) are evaluated negatively. The scale is scored out of a total of 140 points. As the scale score increases, individuals' self-care ability increases. The Cronbach's alpha coefficient for the scale was determined to be 0.89.

Data Collection Study data will be collected by the researcher using face-to-face interviews between May 2025 and June 2025 from women who meet the study criteria and voluntarily agree to participate. Each young woman will be informed about the purpose and content of the study at the first meeting, and verbal and written consent will be obtained from participants who meet the participation criteria and agree to participate. Pre-test data will be collected using a Personal Information Form, the 23-Item Genital Hygiene Behaviors Scale, and the 35-Item Self-Care Abilities Scale. Administration of these tests takes approximately 15 minutes. Post-test data will be collected four weeks after the pre-test data using the Genital Hygiene Behaviors Scale and the Self-Care Abilities Scale using face-to-face interviews.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 24 years of age,
* Agreeing to participate in the study and signing the consent form,
* Having no communication difficulties,
* Completely completing the data collection form.

Exclusion Criteria:

* Taking a health course,
* Being unable to communicate,
* Not being at school during the training period,
* Filling out the data collection form incompletely.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Self-care power will be assessed using the Self-Care Power Scale. The instrument consists of 35 items scored on a 5-point Likert scale ranging from 0 ("does not describe me at all") to 4 ("describes me very well"). The total score ranges from 0 to 140, w | four weeks after the pre-test administration
Change in genital hygiene behavior will be assessed using the Genital Hygiene Behavior Inventory. The scale consists of 23 items scored on a 5-point Likert scale, covering three subdimensions: general hygiene behavior, menstrual hygiene, and awareness of | four weeks after the pre-test administration

IPD SHARING:
Plan to Share IPD: No
"De-identified individual participant data (IPD) will be available from the corresponding author upon reasonable request, solely for academic research purposes, following publication of the article."

REFERENCES:
- [Background] Tiryaki, S., Gezginci, E., & Göktaş, S. (2021). Sağlık Bilimleri Fakültesi Öğrencilerinin Genital Hijyen Davranışlarının Belirlenmesi. İnönü Üniversitesi Sağlık Hizmetleri Meslek Yüksek Okulu Dergisi, 9(2), 510-522. Https://Doi.Org/10.33715/İnonusaglik.843789
- [Background] Pazarözyurt, A., & Özkan, H. (2023). Gebelerin Sağlık Okuryazarlığı İle Öz Bakım Gücü Arasındaki İlişkinin Değerlendirilmesi. Halk Sağlığı Hemşireliği Dergisi, 5(1), 91-102. Https://Doi.Org/10.54061/Jphn.1154752
- [Background] Nahçıvan N. (1994). Geçerlik Ve Güvenirlik ÇALISMASI: ÖZ-BAKIM GÜCÜ Ölçeği'nin TÜRKÇE'YE UYARLANMASI. Florence Nightingale Journal Of Nursing, 33(7), 109-119.
- [Background] Kumral, M. (N.D.). Investigation of the Relationship Between Self-Care Ability, Genital Hygiene Behaviors and Sexually Transmitted Infections among Women of Reproductive Age.
- [Background] Cohen, J. (1988). Statistical Power Analysis For The Behavioral Sciences. (N. E. Edition, Hillsdale, Ed.; 2nd Ed.).
- [Background] Çi̇ftçi̇, M., Demi̇r, R., Sağlık Bilimleri Fakültesi, R., Bölümü, E., Onsekiz Mart Üniversitesi, Ç., Ror Assistant Professor, T., Öğretim Üyesi, D., Bilimleri Fakültesi, S., Ror, T., Author, C., & Sorumlu Yazar, İ. (N.D.). The Effect Of Genital Hygiene Education Given İn The Postpartum Period On Genital Hygiene Behaviors Of Postpartum Women* Doğum Sonu Dönemde Verilen Genital Hijyen Eğitiminin Lohusaların Genital Hijyen Davranışlarına Etkisi*. Https://Doi.Org/10.58252/Artukluhealt